CLINICAL TRIAL: NCT02823899
Title: A Phase I/II Dose-escalation Study to Evaluate Safety, Tolerability and Immunogenicity of '2-dose Primary Series' Single Strain (Hikojima Serotype) Inactivated Oral Cholera Vaccine Formulations (Two Formulations Based on Total O1 LPS Content), in Sequential Age Descending Population of Healthy Adults and Children
Brief Title: Safety and Immunogenicity of Locally Manufactured New (HL-OCV) Oral Cholera Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: MSD Wellcome Trust Hilleman Laboratories Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-16021
Record Dates: First submitted 2016-06-22; First posted 2016-07-06 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2017-01

CONDITIONS: Cholera
Keywords: cholera vaccine; hikojima serotype; randomized trial; immunogenicity
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HL-OCV (Experimental): Pharmaceutical company in Bangladesh is now producing HL-OCV, with technological support from MSD wellcome trust Hilleman pt. ltd, which meets international Good manufacturing practice( GMP) standards and WHO production guidelines.
  Interventions: Biological: HL-OCV
- Shanchol (Active Comparator): The vaccine is manufactured by Shantha Biotechnics in hyderabad, India and is prequalified by the WHO. Shanchol is available in a single dose. This vaccine is used as two dose regimen.
  Interventions: Biological: Shanchol

INTERVENTIONS:
Biological: HL-OCV — Pharmaceutical company in Bangladesh is now producing HL-OCV, with technological support from MSD wellcome trust Hilleman pt. ltd, which meets international Good manufacturing practice( GMP) standards and WHO production guidelines.
  Arms: HL-OCV
Biological: Shanchol — The vaccine is manufactured by Shantha Biotechnics in hyderabad, India and is prequalified by the WHO. Shanchol is available in a single dose. This vaccine is used as two dose regimen.
  Arms: Shanchol

SUMMARY:
Cholera, a rapidly dehydrating watery diarrheal disease transmitted through water or food contaminated with the bacterium, Vibrio cholerae, is a major cause of morbidity and mortality in low income countries like Bangladesh. In our country, Cholera disease burden consists of both cholera outbreaks and endemic cholera comprising at least 300,000 severe cases and 1.2 million infections each year. To combat this situation, Vaccination against cholera has been proved effective both in endemic and epidemic settings. But, the WHO recommended Dukoral and Prequalified Shanchol are quite expensive for our country perspective. Therefore, locally manufactured OCV can improve the cost effectiveness and make it affordable for all. The hypothesis of this proposal is that Locally produced orally administered whole cell inactivated HL-OCV test formulations A and B are safe and immunogenic in adults and children in Bangladesh as compared to ShancholTM. The results of the study will allow us to understand the safety and immunogenicity outcome of the HL-OCV compared to Shanchol vaccine. The total sample size will be 840 healthy participants. 840 healthy participants (360 adults, 240 Children and Adolescent and 240 young children) of 18-45 years, 5- less than 18 years and 1 year to less than 5 years will be enrolled in the study. Children whose parents/guardians give voluntary consent will be enrolled in the study. The investigators will provide 2 dose of vaccine for three groups in 14 days interval. Test formulations will be locally manufactured and the comparator group will get Shanchol. The Investigators propose to collect three blood samples (Day 0, 14 and 28).

DETAILED DESCRIPTION:
Background : Cholera continues to be a major cause of morbidity and mortality in low income countries including Bangladesh. It is estimated that there are at least 300,000 severe cases and over 4,500 deaths in Bangladesh each year1. The overall morbidity for cholera remains high. A global stockpile of OCV has been created by WHO in 2013 for epidemic and outbreak settings30. However, the global demand for the vaccine far exceeds the present supply for both epidemic and also endemic settings3. It can be envisioned that local production of an affordable OCV for high risk population in endemic settings will improve the present scenario in Bangladesh and other countries.

Knowledge gap: The WHO recommends OCV for use in both endemic and epidemic cholera settings4. At present there are two vaccines that are WHO prequalified. These include Dukoral which is registered in Bangladesh and in over 50 countries. However, the disadvantage of use of Dukoral is that its current price is expensive for Bangladesh and other developing countries. In addition, the need for buffer to formulate the vaccine makes it less fieldable for mass vaccination programs.Another whole killed OCV, ShancholTM, which is WHO prequalified, is based on similar bacterial components as Dukoral and licensed in India but not in Bangladesh. Although this vaccine is relatively affordable it may not be sufficiently cost effective for the Government of Bangladesh to implement it in our poor endemic settings. At present, the vaccine is in short supply and will not be able to meet the global demands. In order to increase supply of OCV and make the vaccine more affordable, MSD Wellcome Trust Hilleman Labs. Pvt. Ltd in collaboration with Goteberg University, Sweden has engineered new oral cholera vaccine HL-OCV,consisting of formaldehyde-inactivated recombinant V.cholerae strain ,MS 1568 expressing both Ogawa and Inaba antigens. The vaccine formulation is quantified on total O1 lipopolysaccharide ,LPS content which is matched to that of ShancholTM ,not less than 600 mcg/ml LPS for O1; Formulation A and higher than Shanchol ,not less than 900 mcg/ml LPS for O1; Formulation B. The vaccine technology is transferred to local manufacturer ,INCEPTA in Bangladesh.

Relevance: The study of this locally manufactured new HL-OCV, among children and adults will be able to give us information regarding the safety and immunogenicity of two different formulations of vaccine, based on LPS content. The study will not only identify safe formulation among the two formulation A or B, but will also be able to show superiority of higher LPS formulation in most naive population in children who are 1-5 years of age. Results of the study will be able to identify and select most suitable formulation in Phase II study for licensure in Bangladesh. This study will further pave the way forward for field studies which could establish field efficacy of vaccine compared to existing vaccines in Bangladesh.

Hypothesis : Locally produced orally administered whole cell inactivated HL-OCV test formulations A and B are safe and immunogenic in adults and children in Bangladesh as compared to Shanchol TM.

Objectives: The objective of this study is to determine most safe and immunogenic formulation for new oral cholera vaccine HL-OCV, and comparing with licensed vaccine ShancholTM.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1years to less than 5 years for the younger children group; 5- less than18 years for older children and adolescent group and 18- 45 years (inclusive) for the adult group.
2. Sex: Male, Female, Transgender.
3. Consent: Informed consent from study participants and guardian in case of children along with assent in children 11-17 years (inclusive) of age.
4. Apparently healthy.

Exclusion Criteria:

1. Suffering from diarrhoea or abdominal pain or vomiting in the past 24 hours or diarrhoea lasting for more than 2 weeks in the past 6 months
2. History of taking oral cholera vaccine.
3. History of taking any other live or killed enteric vaccine in the last 8 weeks.
4. History of anaphylaxis or serious vaccine reaction.
5. Currently use of any immunosuppressive or immune-modifying drugs.
6. Receipt of blood or blood products or parenteral immunoglobulin preparation in the past 3 months.
7. Currently on antimicrobial therapy (taking antibiotics within 24 hours during screening and vaccination).
8. Severe malnutrition defined as wt-for-ht z-score <-3.0 with or without oedema.
9. For married females pregnancy or plans to become pregnant during the study period (as determined by verbal screening) will be excluded. In addition, pregnancy test will be done by pregnancy strip test before each day of vaccination (Day 0 and day 14) for married female.
10. Culture positive V. cholerae, ETEC, Salmonella and Shigella in stool.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 840 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with vaccine related reactogenicity as assessed by study personnel. | Within 30 minutes after administration of vaccine
  Number of participants having reactogenicity events will be compared between test group and comparator group
Number of participants with solicited adverse events as assessed by study personnel | Within 7 days after administration of vaccine
  Number of participant having solicited adverse events observed after each dose of vaccination assessed by study personnel through home visit and will be compared between test group and comparator group.
Number of participants with unsolicited adverse event including serious adverse event as assessed by study personnel. | Within 14 days after administration of vaccine.

SECONDARY OUTCOMES:
Number of participant showing seroconversion of vibriocidal antibody against serogroup O1 Inaba | 14 days after administration of vaccine
  Number of participants showing sero-conversion against V. cholerae O1 upon vaccination HL-OCV being tested in comparison with Shanchol TM .
Number of participant showing seroconversion of vibriocidal antibody against serogroup O1 Ogawa. | 14 days after administration of vaccine
  Number of participants showing sero-conversion against V. cholerae O1 upon vaccination HL-OCV being tested in comparison with Shanchol TM .

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, Dr., Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal disease Research,Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with MSD Wellcome Trust Hilleman Laboratories (P) Ltd.

REFERENCES:
- [Result] Ali M, Lopez AL, You YA, Kim YE, Sah B, Maskery B, Clemens J. The global burden of cholera. Bull World Health Organ. 2012 Mar 1;90(3):209-218A. doi: 10.2471/BLT.11.093427. Epub 2012 Jan 24. PMID 22461716
- [Result] Schwartz BS, Harris JB, Khan AI, Larocque RC, Sack DA, Malek MA, Faruque AS, Qadri F, Calderwood SB, Luby SP, Ryan ET. Diarrheal epidemics in Dhaka, Bangladesh, during three consecutive floods: 1988, 1998, and 2004. Am J Trop Med Hyg. 2006 Jun;74(6):1067-73. PMID 16760521
- [Result] Harris JB, LaRocque RC, Chowdhury F, Khan AI, Logvinenko T, Faruque AS, Ryan ET, Qadri F, Calderwood SB. Susceptibility to Vibrio cholerae infection in a cohort of household contacts of patients with cholera in Bangladesh. PLoS Negl Trop Dis. 2008 Apr 9;2(4):e221. doi: 10.1371/journal.pntd.0000221. PMID 18398491
- [Derived] Chowdhury F, Ali Syed K, Akter A, Rahman Bhuiyan T, Tauheed I, Khaton F, Biswas R, Ferdous J, Al Banna H, Ross AG, Mc Millan N, Sharma T, Kanchan V, Pal Singh A, Gill D, Lebens M, Nordqvist S, Holmgren J, Clemens JD, Qadri F. A phase I/II study to evaluate safety, tolerability and immunogenicity of Hillchol(R), an inactivated single Hikojima strain based oral cholera vaccine, in a sequentially age descending population in Bangladesh. Vaccine. 2021 Jul 22;39(32):4450-4457. doi: 10.1016/j.vaccine.2021.06.069. Epub 2021 Jul 1. PMID 34218960